CLINICAL TRIAL: NCT07170540
Title: Cashew Allergy Study in Children: Assessing Desensitization, Efficacy, and Safety (CASCADES Study)
Brief Title: UNC Cashew Sublingual Immunotherapy
Acronym: CASCADES
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Food Allergy Research & Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-2373; G-202401-00621 (Other Grant/Funding Number: Food Allergy Research and Education)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Cashew Nut Allergy; Tree Nut Allergies
Keywords: cashew allergy; tree nut allergy; food allergy; sublingual immunotherapy; SLIT
MeSH Terms: conditions — Nut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cashew SLIT (Active Comparator): Glycerinated cashew extract for sublingual immunotherapy
  Interventions: Drug: Cashew sublingual immunotherapy
- Placebo control (Placebo Comparator): Glycerinated for placebo sublingual immunotherapy
  Interventions: Drug: Placebo sublingual immunotherapy

INTERVENTIONS:
Drug: Cashew sublingual immunotherapy — Glycerinated cashew extract for use in sublingual immunotherapy
  Arms: Cashew SLIT
Drug: Placebo sublingual immunotherapy — Glycerinated saline for placebo sublingual immunotherapy
  Arms: Placebo control

SUMMARY:
The CASCADES study will investigate the safety and efficacy of sublingual immunotherapy (SLIT) for the treatment of cashew allergy in children ages 1-11 years old. Primary efficacy will be assessed after 18 months of cashew SLIT. Lab studies and an oral food challenge after 6 months of cashew SLIT will help determine how quickly cashew SLIT begins to take effect.

DETAILED DESCRIPTION:
The CASCADES study is an 18-month randomized, placebo-controlled trial of cashew sublingual immunotherapy (CASHEW SLIT) in children 1-11 years of age with cashew allergy . Children ages 1-11 years with double-blind placebo-controlled food challenge (DBPCFC) proven allergy to cashew randomized 2:1 to active cashew SLIT or placebo. Participants will undergo a 5-month dose buildup period followed by a DBPCFC at month 6. Participants will then complete an additional 12 months of maintenance cashew SLIT or placebo followed by a DBPCFC at month 18. Safety will be assessed throughout the study. Skin prick testing (SPT), blood sampling, and saliva collection will be performed at baseline and at months 1, 3, 6, 12, and 18 to evaluate for immune biomarker changes.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-11 years at enrollment
* Cashew allergy, with allergy defined as:
* History of clinical reaction to cashew AND cashew-specific IgE >/=0.35 kUA/L AND cashew SPT >/=3 mm
* OR if no prior reaction, cashew-specific IgE >/=5 kUA/L AND cashew SPT >/=3 mm
* Positive Double-Blind Placebo Controlled Food Challenge (DBCPFC) to 443 mg cumulative cashew at enrollment
* If female of child-bearing potential, must have a negative urine or serum pregnancy test
* If female of childbearing potential (defined as females who have reached menarche or who are 12 years or older), must agree to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive methods (barrier methods or oral, injected, or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy) during the treatment period

Exclusion Criteria:

* Inability or unwillingness of a participant and/or parent/legal guardian to give written informed consent and/or assent or comply with the study protocol
* History of severe anaphylaxis to cashew defined as neurological compromise or requiring intubation/mechanical ventilation
* Known oat, wheat, or glycerin allergy
* Poorly controlled or severe asthma/wheezing at screening, defined by at least one of the following criteria:
* Global Initiative for Asthma (GINA) 2024 criteria for uncontrolled asthma
* History of 2 or more systemic corticosteroid courses within 6 months of screening or one course of systemic corticosteroids within 3 months of screening to treat asthma/wheezing
* Prior intubation/mechanical ventilation for asthma/wheezing
* Hospitalization or overnight Emergency Department (ED) visit for asthma/wheezing within 6 months of screening
* Forced expiratory volume in one second (FEV1) <80% of predicted or FEV1/forced vital capacity (FVC) <75%, with or without controller medications (for participants >/= 6 years and older, able to perform spirometry)
* Peak expiratory flow rate (PEFR) <80% of predicted for participants >6 and able to perform peak flow
* Inhaled corticosteroid (ICS) dosing of >500 mcg daily fluticasone (or equivalent ICS)
* Eosinophilic or other inflammatory (e.g., celiac) gastrointestinal disease
* Inability to discontinue antihistamines at least 5 half-lives before scheduled SPT and DBPCFC
* Food immunotherapy such as Oral Immunotherapy (OIT), Sublingual Immunotherapy (SLIT), or Epicutaneous (EPIT) for cashew or pistachio within 6 months of enrollment
* Monoclonal antibodies such as omalizumab (Xolair), dupilumab (Dupixent), benralizumab (Fasenra), mepolizumab (Nucala), or other immunomodulatory therapy within 6 months of enrollment
* Currently on dose escalation of environmental allergen immunotherapy (SCIT or SLIT). Individuals on maintenance allergen immunotherapy can be enrolled
* Participation in any interventional study within the past 3 months
* Pregnant or breastfeeding
* Past or current medical condition or clinical significant laboratory abnormality that, in the opinion of the PI, would make the participant unsafe or otherwise unsuitable for participation in the clinical trial

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Desensitization to cashew at month 18 | 18 months
  Percentage of participants tolerating >/= 1043 mg during cashew DBPCFC at month 18

SECONDARY OUTCOMES:
Full desensitization to cashew at month 18 | 18 months
  Percentage of participants passing the 4043 mg cashew DBPCFC at month 18
Desensitization to cashew at month 6 | 6 months
  Percentage of participants passing the 1043 mg cashew DBPCFC at month 6
Adverse events related to study drug dosing | 18 months
  Percentage of participants reporting adverse events within 2 hours of study drug administration determined by the PI to be possibly or probably associated with study drug dosing.
Change in cashew skin prick testing | Baseline, Months 6 and 18
  Change in SPT wheal to cashew extract
Change in cashew Immunoglobulin E (IgE) | Baseline, Months 6 and 18
  Change in cashew-specific IgE (blood samples)
Change in cashew Immunoglobulin G4 (IgG4) | Baseline, Months 6 and 18
  Change in cashew-specific IgG4 (blood samples)
Change in Cashew-Specific IgG4/IgE Ratio | Baseline, Months 6 and 18
  Change in cashew-specific IgG4/IgE ratio (blood samples)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin H Kim, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.